CLINICAL TRIAL: NCT01034098
Title: Ventilatory Constraint, Breathing Pattern and Ventilatory Responses in Obese Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Li-Ying Wang, School and Graduate Institute of Physical Therapy, National Taiwan University
Other Study IDs: 9461701144
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Obesity; Postmenopausal Women
Keywords: Obesity; Postmenopausal women; Mechanical ventilatory constraints; Dynamic lung volume; Expiratory flow limitation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Post-menopausal women: Post-menopausal women (without hormone replacement therapy)

SUMMARY:
The purpose of this study was to examine the dynamic lung volumes in obese post-menopausal women (without hormone replacement therapy) during exercise and their correlations with dyspnea.

DETAILED DESCRIPTION:
Obesity-related changes in lung volumes have shown to affect breathing mechanisms. During exercise, altered breathing mechanisms increase potential for expiratory flow limitation and compromise exercise capacity. Estrogen and progesterone are potent respiratory stimulants, and their effects in the physiologic regulation of breathing are down-regulated after menopause. Therefore, we theorized that the combined obesity and reduced sex hormone levels after menopause work as a double jeopardy to cause mechanical ventilatory constraint which aggravates dyspnea sensation during exercise, and thus a reduction in exercise capacity. The purpose of this study was to exam the dynamic lung volumes in obese post-menopausal women (without hormone replacement therapy) during exercise and their correlations with dyspnea.

From doctoral referral and advertisement, 24 obese (BMI ≧ 27 kg/m2) and 26 lean post-menopausal women were recruited for the study. Pulmonary function and body composition were measured at rest. A maximal flow volume loop (MFVL) was obtained at baseline. All subjects then performed an incremental exercise test on a cycle ergometer with workload increasing 25 watts every 3 min. During exercise, at each workload, the tidal exercise FV loops were obtained and an inspiratory capacity (IC) maneuver was conducted to assess changes in end-expiratory lung volume (EELV) and end inspiratory lung volume (EILV). Dyspnea and leg fatigue were assessed using the Borg scale. Analysis of variance with repeated measurements was used to test the significance of the mean differences between the two groups during exercise. Linear regression analysis was used to determine whether changes in dynamic lung volumes during exercise were related to changes in Borg scores. Statistical significance was established at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (for at least 1 year)
* Age below 69 y/o
* Not receiving hormone replacement therapy

Exclusion Criteria:

* Cardiopulmonary disease
* Musculoskeletal disease affecting results of maximal exercise test

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women (for at least 1 year) who aged below 69 y/o without hormone replacement therapy
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2005-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Dynamic lung volume: end-expiratory lung volume (EELV), end-inspiratory lung volume (EILV) | At least 1 year post-menopause

SECONDARY OUTCOMES:
Pulmonary function | At least 1 year post-menopause
Breathing pattern | At least 1 year post-menopause
Ventilatory response | At least 1 year post-menopause
Visual analog scale (VAS) for dyspnea and leg fatigue | At least 1 year post-menopause

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Wang, Ph.D., Principal Investigator — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan